CLINICAL TRIAL: NCT02821494
Title: Phase I Study: to Determine the Biological Activity of Two HPV16 E6 Specific Peptides Coupled to Amplivant®, a Toll-like Receptor Ligand in Patients Treated for HPV16-positive Tumors or Premalignant Lesions
Brief Title: Hespecta Vaccination in HPV+ Tumors or Malignant Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leiden University (Other)
Collaborators: ISA Pharmaceuticals (Industry); Dutch Cancer Society (Other); Top Institute Pharma (Other)
Responsible Party: Principal Investigator, HansGelderblom, professor, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HPV16HH01
Record Dates: First submitted 2016-06-02; First posted 2016-07-01 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Tumors or Premalignant Lesions
Keywords: HPV; Vaccination; Immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hespecta (Experimental): Four dose groups of Hespecta
  Interventions: Biological: Hespecta

INTERVENTIONS:
Biological: Hespecta — A dose escalation of Amplivant® conjugated peptide
  Other Names: HPV 16 E6 synthetic peptides (E6 71-95 and E6 127-158)

SUMMARY:
A phase I study to establish the highest safe dose that induces HPV16 E6-specific T-cell responses, using the highly promising novel therapeutic vaccine concept named: Hespecta (HPV E Six Peptide Conjugated To Amplivant®) to induce HPV16 E6-specific T-cell responses.

DETAILED DESCRIPTION:
Human papillomavirus (HPV) has been found to be associated with several types of premalignant lesions and cancer. HPV16 is the far most common HPV type detected in these tumors and premalignant lesions. HPV16 encodes the two tumor-specific oncoproteins E6 and E7. In most humans the virus is cleared. However, in some individuals, infection results in an uncontrolled persistent HPV16 infection that due to expression of the viral oncoproteins E6 and E7 may lead to the formation of malignancies. Moreover, these oncoproteins maintain the malignant state of the transformed cells. The virus-specific interferon-γ (IFNγ)-producing cluster of differentiation 4 (CD4+) helper T cells (Th1 cells) and cluster of differentiation 8 (CD8+) cytotoxic T-lymphocytes (CTL) are able to recognize peptides processed from the highly immunogenic E6 and play a critical role in the elimination and/or control of the virus. Studies in patients with HPV associated tumors showed that the spontaneous HPV-specific T-cell responses, are weak and fail to sufficiently control tumor outgrowth. Preexisting specific T-cell responses against E6 and E7 in patients with HPV related tumors such are associated with better outcome after treatment. Since the HPV16-transformed tumor cells constitutively express the two HPV16 encoded E6 and E7 oncoproteins, these viral antigens are considered to be excellent targets for immunotherapeutic vaccine strategies aiming at reinforcing the tumor-specific T-cell response. Previous vaccination studies showed that the use of our first generation HPV16 synthetic long peptides vaccine (HPV16-SLP) was safe and highly immunogenic in patients with HPV-induced ano-genital lesions. Vaccination of patients with cervical cancer (CxCa) also resulted in the induction of HPV16-specific T-cell responses but the nature and strength of the induced T cell responses was not sufficient for the regression of these tumors. Specifically, it was concluded that the polarization of the T cell response to Th1 (IFNγ-response) was not optimal and a much stronger CD8+ T cell response was required for clinical efficacy. These results initiated the development of new HPV16 vaccination strategies that are able to polarize the induced Th1 response and obtain strong CD8+ T-cell cytotoxicity. One of these developments consists of conjugating two of the HPV16 E6 SLP to Amplivant® a synthetic Toll-like receptor (TLR) 2 ligand. These two peptides cover the most immunodominant regions of the overlapping HPV16-SLP set and contain both Th and CTL epitopes. Peptide conjugated Amplivant® has been selected because it is acknowledged for its capacity to strongly enhance antigen presentation by dendritic cells (DCs), enhance T-cell priming and cause superior induction of effective anti-tumor CTL responses in mouse tumor models, compared to a mixture of free TLR ligand and peptide. In preclinical murine studies, Amplivant®-conjugated SLP showed 10 to 100 times higher bioactivity compared to unconjugated SLP, in terms of induced immune responses. In addition, the quantity and quality of human T-cell responses, and especially the HPV16-specific CD8+ T-cell response, in cancer patients could be markedly enhanced by ex vivo stimulation with Amplivant®-conjugated SLPs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented evidence of HPV16 positive (pre)malignant lesion following standard treatment
2. Patient with a tumor should have no evidence of residual disease based on physical examination at the completion of curative intent therapy
3. At least four weeks and less than twelve weeks after last anti-tumor treatment
4. Willing and able to comply with the protocol and to provide informed consent in accordance with institutional and regulatory guidelines
5. Patients must be 18 years or older.
6. Patients of child-bearing potential should test negative using a serum pregnancy test and agree to utilize effective contraception during the entire treatment and follow-up period of the study (up to 2 months after the last vaccination)
7. Patients must be in good general health and ambulatory, with an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

1. Radiotherapy, chemotherapy or other potentially immunosuppressive therapy administered within 4 weeks prior to the enrolment visit
2. History of an autoimmune disease or other systemic intercurrent disease that might affect the immunocompetence of the patient, or patients receiving immunosuppressive therapy, except for topical application
3. History of a second malignancy except curatively treated low-stage tumors with a histology that can be differentiated from the current tumor or premalignant lesion
4. Receipt of another investigational product within the previous 4 weeks or at any time during the study period.
5. Receipt of prior HPV directed immunotherapy
6. Hematology and biochemistry:

   * Absolute Neutrophil Count (ANC) < 1.5 x 109/L, or platelet count < 100 x 109/L or hemoglobin < 6 mmol/L.
   * Serum (total) bilirubin > 2 x upper normal limit (ULN);
   * Aspartate Aminotransferase (ASAT) or Alanine Aminotransferase (ALAT) > 2.5 x ULN;
   * Alkaline phosphatase levels > 2.5 x ULN;
   * Serum creatinine > ULN or calculated clearance </= 40 mL/min/1.73 m2 for patients with serum creatinine levels above the institutional normal value
7. Human immunodeficiency virus (HIV), chronic hepatitis B or C infection.
8. Any condition that in the opinion of the investigator could interfere with the conduct of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Biological activity of Hespecta | 26 weeks
  Blood samples will be drawn and used in an array of complementary immunological assays to assess the biological activity of Hespecta. Vaccine induced immunity in the different assays is defined if the response after vaccination is at least 3-fold higher than the pre-vaccination response.

SECONDARY OUTCOMES:
Adverse events (AE) according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 26 weeks
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: H. Gelderblom, Prof.dr., Principal Investigator — Leiden University Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Speetjens FM, Welters MJP, Slingerland M, van Poelgeest MIE, de Vos van Steenwijk PJ, Roozen I, Boekestijn S, Loof NM, Zom GG, Valentijn ARPM, Krebber WJ, Meeuwenoord NJ, Janssen CAH, Melief CJM, van der Marel GA, Filippov DV, van der Burg SH, Gelderblom H, Ossendorp F. Intradermal vaccination of HPV-16 E6 synthetic peptides conjugated to an optimized Toll-like receptor 2 ligand shows safety and potent T cell immunogenicity in patients with HPV-16 positive (pre-)malignant lesions. J Immunother Cancer. 2022 Oct;10(10):e005016. doi: 10.1136/jitc-2022-005016. PMID 36261215